CLINICAL TRIAL: NCT05134064
Title: 68Ga-PSMA PET/CT Imaging in Assessment of PCa: Feasibility of Delayed Acquisition on Total-body PET/CT Scanner?
Brief Title: 68Ga-PSMA PET/CT Imaging in Assessment of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yumei Chen, deputy head of the department of nuclear medicine, RenJi Hospital
Other Study IDs: 2018-104
Record Dates: First submitted 2021-11-03; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: PET/CT; Prostate Specific Membrane Antigen; IMAGE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- PCa patients underwent 1 h p.i. PSMA PET/CT imaging and 3 h p.i. PSMA imaging
  Interventions: Device: total-body PET/CT

INTERVENTIONS:
Device: total-body PET/CT — PCa patients who underwent PSMA PET/CT in our clinical center received two-time points scans at 1 h p.i. and 3 h p.i. on a total-body PET/CT scanner.

SUMMARY:
Dual-time point 68Ga-PSMA PET/CT could increase the lesion detection in PCa patients, it remains difficult to perform in clinical practice. The possibility of one-time point 68Ga-PSMA PET/CT imaging could be achieved using a total-body PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* primary staging of pathology-confirmed PCa or evidence of BCR with PSA value > 0.2 ng/ml
* positive 68Ga-PSMA findings
* both standard and delayed scans were performed on the total-body PET/CT

Exclusion Criteria:

* only one scan was performed
* negative PSMA results

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The prospective study consisted of 56 patients for 68Ga-PSMA-11 total-body PET/CT examination between December 2020 and July 2021.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Only one-time point scan is possible for PSMA PET/CT | 8 months
  By the use of total- body PET/CT scanner, the imaging quality between the 1 h p.i. and 3 h p.i. imaging acquisition are compared. And the different lesion detection rates at 3 h p.i. and 1 h p.i. are also discussed. The uptake value differences of all lesions are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No